CLINICAL TRIAL: NCT06823518
Title: Thrive Initiative Domestic and Chlid Abuse Prevention Programming Study
Brief Title: Thrive Initiative Parent-Education Programming Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ryan Chesnut, Assistant Research Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00026099; FA701425C0004 (Other Grant/Funding Number: United States Department of the Air Force)
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-02

CONDITIONS: Child Maltreatment; Parenting; Child Wellbeing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online-Only Thrive Inititaive Parent-Education Programming Condition (Experimental): This arm involves the online-only versions of the Thrive Initiative parent-education programs.
  Interventions: Behavioral: Thrive Initiative Parent-Education Programming
- Hybrid Thrive Initiative Parent-Education Programming Condition (Experimental): This arm involves the hybrid version of the Thrive Initiative parent-education programs. The hybrid version includes the online version and weekly group meetings that can occur in-person or virtually.
  Interventions: Behavioral: Thrive Initiative Parent-Education Programming

INTERVENTIONS:
Behavioral: Thrive Initiative Parent-Education Programming — The Thrive Initiative Parent-Education programs are universal prevention programs designed to support parents as they raise their children. There are four programs that correspond to specific child developmental periods. The programs include: Take Root for parents/caregivers of 0-3-year-old children; Sprout for parents/caregivers of 3-5-year-old children; Grow for parents/caregivers of 5-10-year-old children; and Branch Out for parents/caregivers of 10-18-year-old children. Each program focuses, in developmentally appropriate ways, on three primary dimensions: positive parenting, stress management, and healthy lifestyles. Each program is available in either an online-only format or a hybrid format, which includes group meetings in addition to the online program components.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Thrive Initiative's parent-education program delivery methods by comparing hybrid (i.e., a combination of online and group components) program delivery to online-only program delivery. The Thrive Initiative consists of four, universal parent-education programs that correpsond to specific child developmental periods. These programs inlcude: Take Root for parents/caregivers of 0-3-year-old children; Sprout for parents/caregivers of 3-5-year-old children; Grow for parents/caregivres of 5-10-year-old children; and Branch Out for parents/caregivers of 10-18-year-old children. The effectiveness of delivery method will be examined for each program. Eligible participants for this study will be United States Air Force service members or dependents who are caregivers of a child 0-18 years old. The study will involve randomization to condition meaning that participants will be assigned to the online-only or hybrid program delivery condition by chance.

ELIGIBILITY:
Inclusion Criteria:

* United States Air Force service member or dependent
* Parent/caregiver of a child 0-18 years old
* 18 years of age or older
* Willing to participate in the research study
* Has access to technology that will enable them to receive and respond to various technological aspects of the Thrive Initiative programs and research study
* Able to speak and understand English proficiently
* Able to understand and give consent

Exclusion Criteria:

* Not an United States Air Force service member or dependent
* Not a parent/caregiver of a child 0-18 years old
* 17 years of age or younger
* Unwilling to participate in the research study
* Does not have access to technology that will enable them to receive and respond to various technological aspects of the Thrive Initiative programs and research study
* Unable to speak and understand English proficiently
* Unable to understand and give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ages & Stages Questionnaire: Social-Emotional (2nd Edition) | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of child social-emotional development is administered for the Take Root and Sprout programs. The measure includes five domains (communication, gross motor, fine motor, problem-solving, and personal-social). Scores within each domain range from 0 to 60 with higher scores reflecting typical development.
Mindful Self-Care Scale | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants' self-care strategies, in the domains of physical care, mindful relaxation, and supportive living and work enivronments and schedules, is administered for the Take Root program. Domain scores range from 1 to 4 with higher scores indicating greater engagement in self-care.
National Survey of Early Childhood Health - Discipline Items | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants discipline practices is administered for the Take Root and Sprout programs. Item scores range from 1 to 4 with higher scores reflecting more frequent use of the stated discipline practice.
Parental Stress Scale | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of parenting stress is administered for the Take Root, Sprout, Grow, and Branch Out programs. Scores range from 7 to 35 with higher scores indicating greater stress.
Parenting Sense of Competence Scale | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of parenting efficacy and satisfaction is administered for the Take Root, Sprout, Grow, and Branch Out programs. For the efficacy domain, scores range from 9 to 54. For the satisfaction domain, scores range from 7 to 42. Higher scores indicate greater efficacy and satisfaction.
Positive Behavior Scale | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of positive child behavior, which assesses the domains of social competence, compliance, and autonomy, is administered for the Take Root and Sprout programs. Domain scores range from 1 to 5 with higher scores indicating more positive behavior.
Protective Factors Survey | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of protective factors for child maltreatment, which includes family functioning, emotional support, concrete support, and nurturing and attachment, is administered for the Take Root and Sprout programs. Scores for each factor range from 1 to 7 with higher scores reflecting greater protection.
Co-Viewing Media & Screen Time Recall | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants' co-viewing behavior with their child and their child's screen time is administered for the Sprout program. Participants separately record the amount of time, in minutes and hours, they spend co-viewing media with their child and their child's screen time. The lower bound for the measure is 0, and there is no specific upper bound. Higher scores reflect greater time spent co-viewing media and greater screen time.
Outdoor Time Recall | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of a child's time spent playing outdoors is administered for the Sprout and Grow programs. Participants record, in minutes and hours, the amount of time their child spends playing outside. The lower bound is 0, and there is no specific upper bound. Higher scores reflect greater time spent playing outdoors.
Parenting Scale - Short Form | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of the participants' discipline orientation, which involves the domains of over-reactivity and laxness, is administered for the Sprout and Grow programs. Domain scores range from 1 to 7 with higher scores indicating greater over-reactivity or laxness.
Parenting Young Children Scale | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants' positive parenting practices, which includes the domains of supporting good behavior, setting limits, and proactive parenting, is administered for the Sprout program. Domain scores range from 7 to 49 with higher scores indicating more frequent engagement in positive parenting practices.
Strengths & Difficulties Questionnaire | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of a child's behavior, which includes the domains of conduct problems, hyperactivity/inattention, peer problems, emotional symptoms, and prosocial behavior, is administered for the Sprout, Grow, and Branch Out programs. Domain scores range from 0 to 10. For domains related to externalizing and internalizing behaviors, higher scores indicate more problematic functioning. For the prosocial domain, higher scores indicate greater positive functioning.
Alabama Parenting Questionnaire - 9 | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants' parenting behavior, which assesses the domains of positive parenting, inconsistent discipline, and poor parental monitoring, is administered for the Grow and Branch Out programs. Domain scores range from 1 to 5 with higher scores reflecting more frequent positive parenting, inconsistent discipline, and poor parental monitoring.
Feeding Practices & Structure Questionnaire | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of the feeding behaviors and environment participants use with their children is administered for the Grow program. The specific domains assessed include using food as a reward for behavior and using rewards to encourage eating. Domain scores range from 1 to 5 with higher scores indicating more problematic feeding practices.
Healthy Habits Index | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants encouragement and support of healthy habits in their children is administered for the Grow program. Scores ranges from 1 to 5 with higher scores reflecting greater engagement in healthy behaviors.
Interpersonal Mindfulness in Parenting Scale | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants use of mindfulness in their parenting is administered for the Grow program. Scores range from 1 to 5 with higher scores indicating greater incorporation of mindful practices in participants' parenting approach.
Parental Emotional Styles Questionnaire | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants use of emotion regulation orientation is administered for the Grow program. Scores range from 1 to 5 with higher scores reflecting an emotion-coaching, as opposed to an emotion-avoidant, parenting style.
Socialization of Coping Questionnaire | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of participants encouragement of their child's development of different coping strategies, which includes the domains of primary control engagement and cognitive restructuring, is administered for the Grow program. Domain scores range from 1 to 5 with higher scores reflecting greater encouragment of the indicated coping strategy.
Family Assessment Device - General Functioning | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of general family functioning is administered for the Branch Out program. Scores range from 1 to 4 with higher scores reflecting worse family functioning.
Parent-Adolescent Communication Scale | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of parent-adolescent communication, which assesses the domains of open and problematic communication, is administered for the Branch Out program. Domain scores range from 1 to 5 with higher scores in each domain indicating more open and problematic communication patterns.
Targeted Parent-Child Communication about Substances Scale | Baseline (2 weeks before intervention start), up to 6 weeks after intervention start, and 6 months after intervention end
  This measure of the participants communication with their child about substances is administered for the Branch Out program. Scores range from 1 to 5 with higher scores indicating more explicit or intentional communication about substance use.

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire-8 | Up to 6 weeks after intervention start
  This measure of participant satisfaction is adminstered for the Take Root, Sprout, Grow, and Branch Out programs. Scores range from 8 to 32 with higher scores reflecting greater satisfaction.
Program Noncompletion Reason(s) Survey | Up to 6 weeks after intervention start
  This measure of program participation barriers is administered for Take Root, Sprout, Grow, and Branch Out. Participants select the most appropriate barriers from the list provided, and they are given the option to write in additional barriers not listed.

OTHER OUTCOMES:
Demographic Survey | Baseline (2 weeks before intervention start)
  This measure of participants' demographic and contextual characteristics is administered for Take Root, Sprout, Grow, and Branch Out.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Perkins, PhD, Principal Investigator — The Pennsylvania State University; Ryan P Chesnut, PhD, Principal Investigator — The Pennsylvania State University

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared per the guidance received from the United States Department of the Air Force.